CLINICAL TRIAL: NCT00392067
Title: LEO19123 Cream in the Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEO19123-C21
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2007-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — calcipotriene

INTERVENTIONS:
Drug: Calcipotriol and LEO80122 (LEO19123 cream)

SUMMARY:
To compare the efficacy and safety of two different dose combinations of LEO19123 (calcipotriol and LEO80122) with LEO19123 cream vehicle for 3 weeks in the treatment of patients with atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of atopic dermatitis according to Hanifin and Rajka
* The score of erythema, induration/papulation, excoriation and lichenification, four of the five clinical signs in the Total Severity Score, should at least correspond to moderate involvement, i.e. severity greater than or equal to 2, at Visit 1
* Treatment area amenable to topical treatment
* Attending a hospital outpatient clinic or the private practice of a dermatologist
* Following verbal and written information about the trial, the patient must provide signed and dated informed consent before any study related activity is carried out, including activities relating to washout period
* Males between 18-50 years

Exclusion Criteria:

* Systemic treatment with immunosuppressive drugs (e.g. methotrexate, cyclosporine, azathioprine) or corticosteroids within 4 weeks prior to randomisation. (Inhaled or intranasal steroids for asthma or rhinitis may be used)
* PUVA or UVB therapy within 4 weeks prior to randomisation
* Topical treatment with immunomodulators (pimecrolimus, tacrolimus) or corticosteroids from WHO groups III or IV within 2 weeks prior to randomisation
* Other topical therapy on the treatment area (except for the use of emollient on the entire body and use of hydrocortisone cream 1% on AD lesions on head and neck) within 1 week prior to randomisation
* Use of any other kind of treatment (drug, non-drug) for AD during the study except for the use of: - Investigational product on trunk and limbs lesions only during the treatment phase - Hydrocortisone cream 1% on head and neck lesions - Emollient on the entire body
* Use of anti-histamines during the study
* Current diagnosis of exfoliative erythrodermia
* Clinical infection (impetiginised atopic dermatitis) on the treatment area
* Planned exposure to amount of sun or ultraviolet light during the study that may affect atopic dermatitis
* Known or suspected hypersensitivity to component(s) of the investigational product
* Known or suspected severe renal insufficiency or severe hepatic disorders
* Patients with history/signs/symptoms suggestive of an abnormality of calcium homeostasis associated with clinically significant hypercalcaemia
* Patients with history of cancer including skin cancer
* Patients with history of an immunocompromised disease (e.g. lymphoma, HIV, Wiskott-Aldrich Syndrome)
* Current participation in any other interventional clinical trial
* Patients who have received treatment with any non-marketed drug substance (i.e. an agent which has not yet been made available for clinical use following registration) within 4 weeks prior to randomisation
* Previously randomised in this study
* Patients known or suspected of not being able to comply with a trial protocol (e.g. alcoholism, drug dependency, or psychotic state)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2006-10; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Proof of concept

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Thestrup-Pedersen, MD, Principal Investigator — Hudklinikken
Locations (4):
- Clinique Dermatologique Maizerets, Québec, Quebec, Canada
- Hudklinikken, Nykøbing Falster, Denmark
- Helsinki University Central Hospital, Helsinki, Finland
- Manchester Royal Infirmary, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No